CLINICAL TRIAL: NCT00265655
Title: Phase II of Oral Satraplatin in Patients With Metastatic Breast Cancer (MBC)
Brief Title: Satraplatin for Patients With Metastatic Breast Cancer (MBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 05-021
Record Dates: First submitted 2005-12-01; First posted 2005-12-15 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — satraplatin

INTERVENTIONS:
Drug: Satraplatin — Patients will receive 80mg/m2 Satraplatin on Days 1-5 of Cycles 1 and 2. A cycle consists of 21 days.

SUMMARY:
To determine the objective response rate (ORR) of oral satraplatin in patients with Metastatic Breast Cancer.

DETAILED DESCRIPTION:
This is a Phase II open label, nonrandomized study for patients with metastatic breast cancer.

WHAT IS SATRAPLATIN:

Satraplatin is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally.

ELIGIBILITY:
1. Has cytologically or pathologically confirmed breast cancer that is metastatic
2. Must have had prior HerceptinÒ therapy if patient has HER2+ (overexpressing) breast cancer. HER2 is considered overexpressed if it is 3+ by IHC or if the gene is amplified by Flourescence in situ hybridization (FISH)
3. Has had no more than 1 prior chemotherapy regimen for MBC
4. Has had no prior platinum-based therapy
5. Has an ECOG Performance Status (PS) 0-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To determine the objective response rate (ORR) of oral satraplatin in patients with metastatic breast cancer | 1 year

SECONDARY OUTCOMES:
To determine duration of response | 6 weeks
To determine progression-free survival (PFS) | 1 year
To determine 1-year survival | 1 year
To evaluate the toxicities of satraplatin in MBC patients | 6 weeks
In patients with nonmeasurable MBC, to assess the clinical utility of serum CA27.29 (or CA15.3) and circulating tumor cells as predictors of time to disease progression | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, MD, Principal Investigator — US Oncology
Locations (1):
- US Oncology, Dallas, Texas, United States